CLINICAL TRIAL: NCT03552809
Title: Clinical Evaluation of Postoperative Healing After Conventional And Laser Assisted Frenectomy Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cetinkaya et al.
Record Dates: First submitted 2018-03-31; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Frenulum; Hypertrophy, Lip
MeSH Terms: conditions — Hypertrophy; Lymphoid Interstitial Pneumonia | interventions — Lasers, Semiconductor

ARMS (3):
- Conventional Frenectomy (Active Comparator): For the conventional surgery, after application of local infiltration anesthesia of articaine HCL associated with epinephrine 1:100,000, the frenulum was grasped with a straight haemostat inserted into the depth of the vestibule; the tissue adjacent to the upper and lower surfaces of the haemostat was incised with a no.15 scalpel. After the diamond shaped resected portion of the frenulum was removed with the haemostat, muscle dilatations were excised on the submucosa of the lateral walls of the cavity. Horizontal incision was made on the periosteum with the help of a scalpel following the procedure. At the end of the operation, the wound was closed with absorbable sutures (4-0, Pegelak®, Doğsan Turkey).
  Interventions: Procedure: Conventional Frenectomy Operation
- Diode Laser Frenectomy (Experimental): For the laser frenectomy, a diode laser device (λ = 810 nm, W: 4, GIGA Cheese II, China) was used to perform the procedure. The procedure was performed under local infiltration anesthesia with articaine HCL associated with epinephrine 1:100,000. The frenlum was held by a haemostat inserted into the depth of the vestibule while laser energy was applied to the upper and lower parts of the frenulum adjacent to the haemostat via a fibre tip (400 µm diameter, plain-ended, optical ﬁbre). The laser was carefully applied to the tissue and care was taken to avoid local necrosis of the periosteum or any bone structure.Following the bleeding control, the wound site was left to secondary healing. No sutures were necessary after procedure.
  Interventions: Device: Gigaa Cheese 810 nm Diode Laser
- Laser Frenectomy with Incision (Experimental): For the laser frenectomy, a diode laser device (λ = 810 nm, W: 4, GIGA Cheese II, China) was used to perform the procedure. The procedure was performed under local infiltration anesthesia with articaine HCL associated with epinephrine 1:100,000. The frenulum was held by a haemostat inserted into the depth of the vestibule while laser energy was applied to the upper and lower parts of the frenulum adjacent to the haemostat via a fibre tip (400 µm diameter, plain-ended, optical ﬁbre). The laser was carefully applied to the tissue and care was taken to avoid local necrosis of the periosteum. Horizontal incision was made on the periosteum with the help of a scalpel, additionally. No sutures were necessary after procedure.
  Interventions: Device: Gigaa Cheese 810 nm Diode Laser

INTERVENTIONS:
Device: Gigaa Cheese 810 nm Diode Laser — Diode Laser assisted frenectomy operation.
  Arms: Diode Laser Frenectomy; Laser Frenectomy with Incision
Procedure: Conventional Frenectomy Operation — Frenectomy operation performed by surgical blades with suturing.
  Arms: Conventional Frenectomy

SUMMARY:
The aim of this randomized controlled parallel-designed study was to evaluate clinical healing and patient comfort after conventional and diode laser assisted frenectomy operations in case of high papillary frenulum attachment. Forty-eight patients with high papillary frenulum attachments were included in the study. Patients were randomly divided into three groups; conventional frenectomy operation (Group C), frenectomy operation using diode laser (Group L) and diode laser asissted frenectomy with horizontal incision on the periosteum (Group L+P). Postoperative pain, difficulty in speaking and eating scores were assessed postoperative 3 hours and 1, 7, 14, 21 and 45 days using Visual Analogue Scale (VAS). Evaluation of epithelialization of the wound surface was carried out via hydrogen peroxide to the surface using a dental injector at postoperative 7, 14, 21 and 45 days. Plaque index, gingival index, bleeding on probing and probing depth were assessed at baseline and postoperative 7, 14, 21 and 45 days. All data were compared between groups and within each group.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy, nonsmoker, aged between 18 and 65, high papillary frenulum attachment diagnosed according to Mirko et al (Mirko et al, 1974), not received any periodontal treatment within the last 3 months, presence of at least central, lateral incisors and canines at the upper jaw, and consent to participate in the study.

Exclusion Criteria:

* Any systemic disease that might interfere with the prognosis of periodontal disease (i.e., diabetes mellitus, HIV infection), smoking, antibiotics, anti-inflammatory drugs or any other medication taken within the last 6 months that might affect the outcome of the study, any physical limitations or restrictions that might preclude normal oral hygiene procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Change | Postoperative pain, difficulty during speaking and eating scores were assessed on postoperative 3 hours and 1, 7, 14, 21 and 45 days.
  Postoperative pain during eating and speaking will be evaluate via visual analog scale (VAS).Visual Analogue Scale (VAS) was used to evaluate pain, discomfort during speaking and chewing. VAS consisted of a horizontal line with a range of numbers from '0' to '10' of which '0' means 'no pain' and '10' means unbearable pain.